CLINICAL TRIAL: NCT01701908
Title: Postoperative Pulmonary Complications in Major Abdominal Surgery: a Multicenter Prospective Observational Study
Brief Title: Postoperative Pulmonary Complications in Major Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: University of Udine (Other)
Responsible Party: Principal Investigator, Giorgio Della Rocca, MD, Principal Investigator, University of Udine
Other Study IDs: PPC01; NCT01914328 (obsolete NCT alias)
Record Dates: First submitted 2012-09-30; First posted 2012-10-05 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Pulmonary Complications
Keywords: PPCs; abdominal surgery; postoperative infections; postoperative residual curarization; tracheal re-intubation; mortality; ICU stay
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Incidence of Postoperative Pulmonary Complications (PPCs) varies from 2% to 19%, according to the population under examination and the criteria used to define pulmonary complications. There is no univocal definition of PPCs. Usually physicians associate atelectasis, respiratory insufficiency, pneumonia, bronchospasm, necessity to reintubate. Moreover the evaluation of risk factors has become difficult.

The endpoint of this study is to determine the actual incidence of respiratory postoperative complications in patients undergoing general anesthesia for major abdominal surgery (general surgery, gynecology, urology).

This is an observational, descriptive, prospective, multicentric study. Investigators are going to enroll all the patients matching the inclusion criteria and follow them until discharge (clinical phase). Then they will be followed up until one year later.

DETAILED DESCRIPTION:
INTRODUCTION Pulmonary Postoperative Complications (PPCs) are among the most common causes of adverse events in the perioperative period and can determine a significant increase of mortality risk in hospitalization time.

Incidence of PPCs varies from 2% to 19%, according to the population under examination and the criteria used to define pulmonary complications. There is no univocal definition of PPCs. Usually physicians associate atelectasis, respiratory insufficiency, pneumonia, bronchospasm, necessity of tracheal reintubation. Moreover, the evaluation of risk factors is becoming increasingly difficult. Many aspects linked to the patient's conditions and postoperative anesthesiologic management have been demonstrated to influence the risk of developing PPCs. (with the endorsement of European Society of Anesthesiology) proposed a risk index based on seven perioperative parameters to predict PPCs probability.

Furthermore, patients who survive after pulmonary complications will still suffer from functional reductions and are at risk of having a decrease in medium and long-term survival.

PRIMARY END POINT To determine the actual incidence of respiratory postoperative complications in patients undergoing elective general anesthesia for major abdominal surgery (general surgery, urology, gynecology).

Respiratory complications are: pneumonia, respiratory insufficiency, pleural effusion, pneumothorax, atelectasis, ab ingestis pneumonia, necessity of oxygen supply, non invasive mechanical ventilation (NIMV) or tracheal reintubation.

SECONDARY END POINTS

To determine:

* postoperative pulmonary complications rate in general, gynecology and urology
* length of hospital stay
* unplanned postoperative Intensive care unit (ICU) admission and ICU length of stay
* postoperative incidence of tracheal reintubation
* postoperative incidence of infections
* postoperative incidence of PostOperative Residual Curarization (PORC)
* postoperative incidence of cardiovascular complications
* postoperative mortality (in-hospital, 30, 60 days and one year later)

Duration of the clinical phase: hospitalization (data collection: two hours after discharge from the operating room, then from the first, up to the fifth postoperative day and on the day of hospital discharge) Duration of follow-up after hospitalization (follow up period): 30 days - 60 days - 1 year.

RECRUITMENT AND MONITORING PROCEDURES All patients scheduled for elective major abdominal surgery, urologic surgery or major gynecological surgery under general anaesthesia will be enrolled in this study.

Patients will be enrolled over a 15 days period, after that, if the sample would be too small, another 15 days enrollment period will be repeated.

During the preoperative evaluation, the anesthesiologist will expose the study protocol to all patients who will match the inclusion criteria. The informed consent will be obtained.

Patients will be monitored in the postoperative period and will receive, standard postoperative care, as directed by the clinical teams and if indicated, antibiotics, diuretics, oxygen therapy and every therapy according to the underlying disease. Medical and nursing staff will monitor peripheral oxygen saturation in the origin ward.

In every center a researcher will evaluate the enrolled patients daily, checking for peripheral oxygen saturation, arterial pressure, heart rate, respiratory rate, body temperature and pain assessment (NRS scale).

Patient's clinical status until the hospital discharge will be reported on case report forms (CRFs). Every intraoperative parameter (like drugs used, the need of blood transfusion, fluid management and fluid balance at the end of surgery) will be recorded.

Treatments and therapy will be continued according to clinicians decision and will be recorded in the CRF.

The decision to start an oxygen therapy or a ventilatory support (invasive or non-invasive) or to admit the patient to the ICU will be taken by clinicians of every single participating center according to their guidelines.

Every device used, with oxygen flow values, FiO2, PEEP and ventilation mode (assisted/mechanical) will be noted in the CRF..

Anesthesiologist will evaluate all the patients two hours after their return in the ward, and from the first to the fifth postoperative day. Anesthesiologists will be also on-call by the attending physician or the nursing staff every time patient's clinical conditions will need it.

Every patient will be followed (and will be enrolled in the study) until hospital discharge. Date of discharge will be noted in the CRF.

Moreover every enrolled patient will be followed-up at 30, 60 days and a year after hospital discharge, to verify the patients health status and to evaluate the incidence of re-hospitalization and mortality.

DATA COLLECTION:

A form divided in three sections (pre/intra/postoperative period) will be used for data collection. Data will be collected on paper support and then entered in an electronic CRF.

Data will be anonymous. Every patient will be identified by a six number code: first three (from left to right) identify the participating center, the others identify the sequential number of enrollment.

The data insertion will be done by the investigators of every participating center, using personal username and password.

Data will be sent to the coordinator center where the data cleaning will be completed and statistical analysis.

Every center will store its own paper CRF.

In the preoperative section will be recorded the patient's data about:

age, weight, height, sex; comorbidities (neurological, cardiovascular, metabolic, renal, muscular-skeletal) respiratory history positive for: previous pleuro-parenchymal diseases in the 30 days before surgery, previous chest, pleural or lung surgery, presence of pleural effusion; history of cigarettes smoking: active smoker; history of alcohol abuse; active cancer (excluding the diagnosis for surgery); SpO2, PaO2, PaO2/FiO2, PaCO2 when available; white cell number, hemoglobin and preoperative creatinine; ASA class; presence of nasogastric tube before surgery; presence of urinary catheter before surgery; blood products transfusion before surgery.

In the intraoperative section will be recorded the patient's data about:

type of surgery; type of anaesthesia (TIVA, balanced); type of analgesia (intravenous, epidural, perineural block); preoperative antibiotic prophylaxis; blood products transfusion; intraoperative fluid management (crystalloids Vs colloids, mL/Kg/h); type of ventilation (PCV/VCV); ventilation parameters (TV, Pins, PEEP, RR, FiO2); recruitment maneuvers (yes/no) (manuals, pressure controlled); intraoperative ventilatory problems ( (SpO2 < 90%, PaO2/FiO2 < 300, PaCO2 > 45 mmHg, increase of airways pressure over than 30 cmH2O, bronchospasm, needs of TV> 10 mL/Kg); hemorrhage or need of blood products transfusion; cardiovascular problems (hypotension, tachycardia, bradycardia, arrhythmia) and use of cardio/vasoactive drugs;

* length of surgery;
* use of qualitative or quantitative (TOF Watch) neuromuscular transmission monitoring systems use of neostigmine or sugammadex
* Final TOF ratio

In the postoperative section will be recorded the following data:

pain score at discharge from the operating room and up to the fifth postoperative day; needs of blood products transfusion in the postoperative period; stay of nasogastric tube;

* stay of urinary catheter;
* postoperative respiratory complications;
* postoperative non-respiratory complications (cardiovascular, renal, surgical, infections)
* needs of re-intubation in the postoperative period;
* needs of ventilatory support (non invasive ventilation, invasive ventilation) in the postoperative period; needs of ICU admission (planned, unplanned, cause, length of ICU stay); length of hospital stay; 30, 60 days and 1 year mortality (specify the cause).

STATISTICAL PLANS

Investigators are going to enroll 1500 patients undergoing elective major abdominal surgery, in a period of 15 days. It will be possible to add 15 extra days. On the basis of works published by Squadrone et. al.[11] (16%), Lawrence et.al. [17] (4,5%), Hall et. al. [18] (15%), Mitchell et.al. [19] (11%) and Canet et. al. (7,2%) [10], the hypothesis was that the incidence of primary outcome will be 7%.

The sample size has been calculated using alpha = 0,05 (2-tailed test) and CI of 95%.

The result of this calculation is a sample size of 1422. Investigators decided to enroll 1500 patients because this way our population will be heterogeneous and because of possible deviations from the protocol.

The statistic analysis will include:

* descriptive statistics of all the collected data (average, median, standard deviation, interquartile range, minimum and maximum for the continuous variables; relative and absolute frequency for the qualitative variables
* interdependence between two or more variables (if present)
* Statistic comparison between continuous variables, using t-Student test (if the variable has a normal distribution) or non-parametric tests.
* Comparison between qualitative variables, using Chi-square test
* Odds ratio
* Logistic regression
* The study will include the possibility to perform non-planned analyses, if useful.

The data will be saved on an electronic support and analyzed with SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Ability to provide informed consent
* Elective surgery
* Laparotomic or laparoscopic major abdominal surgery
* Major urological surgery (performed under general anesthesia)
* Major gynecological surgery (performed under general anesthesia)

Exclusion Criteria:

* Patients undergoing urgent or emergent surgery
* Patients undergoing: vascular, thoracic ,cardiac surgery, neurosurgery, obstetrics procedures and transplantation surgery
* Patients with chronic neuro-muscular junction disorders
* Immunocompromised or immunodepressed patients
* Patients with chronic or acute respiratory disease (acute respiratory infection, bronchial asthma, chronic obstructive pulmonary disease, sleep apnea syndrome)
* Patients with preoperative mechanical ventilation
* Patients with preoperative SpO2 <90%, PaO2 <60 mmHg (FiO2 0.21), or a PaO2/FiO2 ratio <300, or PaCO2 >45 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1500 patients undergoing elective major abdominal surgery, urologic surgery or major gynecological surgery under general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 1542 (Actual)
Dates: Start 2013-04-17 (Actual); Primary Completion 2014-06-05 (Actual); Study Completion 2015-06-08 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications rate | From surgery to hospital discharge (an average of 10 days)
  Complications are: respiratory infection, postoperative respiratory failure, pleural effusion, pneumothorax, atelectasis, aspiration pneumonia, bronchospasm, need of oxygen supplementation or noninvasive ventilatory support or unplanned urgent re-intubation

SECONDARY OUTCOMES:
Postoperative pulmonary complications rate in general, gynecology and urology | From surgery to hospital discharge (an average of 10 days)
  Pulmonary complications among different type of surgery
Mortality rate after surgery | Up to 1 year after surgery
  Incidence of mortality after surgery in patients with or without postoperative pulmonary complications
Length of hospital stay | From surgery to hospital discharge (an average of 10 days)
  Duration of hospital stay after surgery
Unplanned postoperative Intensive care unit (ICU) admission | From surgery to hospital discharge (an average of 10 days)
  Unplanned ICU admission after surgery
Intensive care unit length of stay | From surgery to hospital discharge (an average of 10 days)
  Duration of ICU stay
Postoperative incidence of tracheal re-intubation | From surgery to hospital discharge (an average of 10 days)
  Re-intubation rate after discharge from the operating room or after ICU discharge
Postoperative incidence of infections | From surgery to hospital discharge (an average of 10 days)
  Occurrence of pneumonia, surgical site infection and any other infections
Postoperative incidence of cardiovascular complications | From surgery to hospital discharge (an average of 10 days)
  Cardiovascular complications: arrhythmias, acute coronary syndrome, mycardial infarction, acute congestive heart failure
Postoperative incidence of PostOperative Residual Curarization (PORC) | Up to 3 hours after extubation
  PORC defined as: train-of-four ratio < 0.9 after extubation or need for reversal drug fo neuromuscular blocking agent after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Della Rocca, Professor, Principal Investigator — University of Udine
Locations (40):
- Italy (40):
  - Ospedale Grassi, Ostia Antica, Rome
  - Istituto di Candiolo, Candiolo, Torino
  - S. Valentino Hospital, Montebelluna, Treviso
  - AO Santa Maria della Misericordia, Udine, UD
  - University of Verona, Bussolengo, Verona
  - Ospedali Riuniti, Ancona
  - Cardinal Massaia Hospital, Asti
  - Irccs Cro, Aviano
  - Policlinico di Bari Ospedale Giovanni XXIII, Bari
  - Ospedale Rummo, Benevento
  - ASST Papa Giovanni XXIII, Bergamo
  - S.Orsola-Malpighi Hospital, Bologna
  - Spedali Civili, Brescia
  - Ospedale Versilia, Camaiore
  - ASST Lariana, Como
  - ASST Cremona, Cremona
  - ASO S Croce e Carle, Cuneo
  - Azienda Ospedaliero-Universitaria, Ferrara
  - Mugello Hospital, Florence
  - S. Maria Nuova Hospital, Florence
  - University of Foggia, Foggia
  - Presidio Ospedaliero Sora, Frosinone
  - IRCCS San Martino, Genova
  - Fazzi Hospital, Lecce
  - Ospedale Provinciale di Macerata, Macerata
  - IRCCS Fondazione Istituto Nazionale dei Tumori, Milan
  - IRCCS S. Raffaele, Milano, Milan
  - Azienda Ospedaliero Universitaria Vanvitelli, Naples
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Naples
  - Ospedale Monaldi, Naples
  - Federico II Hospital, Napoli
  - Nuovo Santa Chiara Hospital, Pisa
  - Irccs Cro, Potenza
  - Azienda USL IRCCS, Reggio Emilia
  - Umberto I, "Sapienza", University of Rome, Rome
  - Catholic University Hospital A. Gemelli, Rome
  - Campus Bio-medico Foundation, Rome
  - Università Cattolica del Sacro Cuore, Rome
  - Ospedale S Chiara, Trento
  - OC San Bortolo, Vicenza

REFERENCES:
- [Background] Smetana GW. Preoperative pulmonary evaluation. N Engl J Med. 1999 Mar 25;340(12):937-44. doi: 10.1056/NEJM199903253401207. No abstract available. PMID 10089188
- [Background] Smetana GW, Lawrence VA, Cornell JE; American College of Physicians. Preoperative pulmonary risk stratification for noncardiothoracic surgery: systematic review for the American College of Physicians. Ann Intern Med. 2006 Apr 18;144(8):581-95. doi: 10.7326/0003-4819-144-8-200604180-00009. PMID 16618956
- [Background] Fleischmann KE, Goldman L, Young B, Lee TH. Association between cardiac and noncardiac complications in patients undergoing noncardiac surgery: outcomes and effects on length of stay. Am J Med. 2003 Nov;115(7):515-20. doi: 10.1016/s0002-9343(03)00474-1. PMID 14599629
- [Background] Khuri SF, Henderson WG, DePalma RG, Mosca C, Healey NA, Kumbhani DJ; Participants in the VA National Surgical Quality Improvement Program. Determinants of long-term survival after major surgery and the adverse effect of postoperative complications. Ann Surg. 2005 Sep;242(3):326-41; discussion 341-3. doi: 10.1097/01.sla.0000179621.33268.83. PMID 16135919
- [Background] Fisher BW, Majumdar SR, McAlister FA. Predicting pulmonary complications after nonthoracic surgery: a systematic review of blinded studies. Am J Med. 2002 Feb 15;112(3):219-25. doi: 10.1016/s0002-9343(01)01082-8. PMID 11893349
- [Background] Antonelli M, Conti G, Bufi M, Costa MG, Lappa A, Rocco M, Gasparetto A, Meduri GU. Noninvasive ventilation for treatment of acute respiratory failure in patients undergoing solid organ transplantation: a randomized trial. JAMA. 2000 Jan 12;283(2):235-41. doi: 10.1001/jama.283.2.235. PMID 10634340
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Early goal-directed therapy after major surgery reduces complications and duration of hospital stay. A randomised, controlled trial [ISRCTN38797445]. Crit Care. 2005;9(6):R687-93. doi: 10.1186/cc3887. Epub 2005 Nov 8. PMID 16356219
- [Background] Brooks-Brunn JA. Predictors of postoperative pulmonary complications following abdominal surgery. Chest. 1997 Mar;111(3):564-71. doi: 10.1378/chest.111.3.564. PMID 9118688
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Dimick JB, Pronovost PJ, Cowan JA Jr, Lipsett PA, Stanley JC, Upchurch GR Jr. Variation in postoperative complication rates after high-risk surgery in the United States. Surgery. 2003 Oct;134(4):534-40; discussion 540-1. doi: 10.1016/s0039-6060(03)00273-3. PMID 14605612
- [Background] McAlister FA, Bertsch K, Man J, Bradley J, Jacka M. Incidence of and risk factors for pulmonary complications after nonthoracic surgery. Am J Respir Crit Care Med. 2005 Mar 1;171(5):514-7. doi: 10.1164/rccm.200408-1069OC. Epub 2004 Nov 24. PMID 15563632
- [Background] Gupta H, Gupta PK, Fang X, Miller WJ, Cemaj S, Forse RA, Morrow LE. Development and validation of a risk calculator predicting postoperative respiratory failure. Chest. 2011 Nov;140(5):1207-1215. doi: 10.1378/chest.11-0466. Epub 2011 Jul 14. PMID 21757571
- [Background] Ware LB, Matthay MA. The acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1334-49. doi: 10.1056/NEJM200005043421806. No abstract available. PMID 10793167
- [Background] Squadrone V, Coha M, Cerutti E, Schellino MM, Biolino P, Occella P, Belloni G, Vilianis G, Fiore G, Cavallo F, Ranieri VM; Piedmont Intensive Care Units Network (PICUN). Continuous positive airway pressure for treatment of postoperative hypoxemia: a randomized controlled trial. JAMA. 2005 Feb 2;293(5):589-95. doi: 10.1001/jama.293.5.589. PMID 15687314
- [Background] Lawrence VA, Dhanda R, Hilsenbeck SG, Page CP. Risk of pulmonary complications after elective abdominal surgery. Chest. 1996 Sep;110(3):744-50. doi: 10.1378/chest.110.3.744. PMID 8797421
- [Background] Hall JC, Tarala RA, Hall JL. Respiratory insufficiency after abdominal surgery. Respirology. 1996 Jun;1(2):133-8. doi: 10.1111/j.1440-1843.1996.tb00022.x. PMID 9434329
- [Background] Mitchell CK, Smoger SH, Pfeifer MP, Vogel RL, Pandit MK, Donnelly PJ, Garrison RN, Rothschild MA. Multivariate analysis of factors associated with postoperative pulmonary complications following general elective surgery. Arch Surg. 1998 Feb;133(2):194-8. doi: 10.1001/archsurg.133.2.194. PMID 9484734